CLINICAL TRIAL: NCT00004346
Title: Effects of Diet and Medication in Patients With Cerebrotendinous Xanthomatosis (CTX)
Brief Title: Phase II Study of Cholesterol- and Cholestanol-Free Diet, Lovastatin, and Chenodeoxycholic Acid for Cerebrotendinous Xanthomatosis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: Oregon Health and Science University (Other)
Purpose: Treatment
Other Study IDs: NCRR-M01RR00334-0067; OHSU-4008
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Cerebrotendinous Xanthomatosis
Keywords: cerebrotendinous xanthomatosis; inborn errors of metabolism; rare disease
MeSH Terms: conditions — Xanthomatosis, Cerebrotendinous; Metabolism, Inborn Errors; Rare Diseases | interventions — Chenodeoxycholic Acid; Lovastatin

INTERVENTIONS:
Drug: chenodeoxycholic acid
Drug: lovastatin

SUMMARY:
OBJECTIVES: I. Assess the biosynthesis of cholesterol and cholestanol, and measure the turnover of individual sterols and bile acids in patients with cerebrotendinous xanthomatosis before and after a cholesterol- and cholestanol-free diet.

II. Assess the biosynthesis of cholesterol and cholestanol, and measure the turnover of individual sterols and bile acids in these patients before and after lovastatin and chenodeoxycholic acid.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Following a 2-week baseline assessment, patients participate in a feeding study for up to 3 weeks. The diet is free of cholesterol and cholestanol.

For the next 4 weeks, patients return to their typical diet and are medicated with daily lovastatin and chenodeoxycholic acid.

The feeding study is repeated for an additional 3 weeks, with the patient taking either lovastatin or chenodeoxycholic acid.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA: Cerebrotendinous xanthomatosis

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5
Dates: Start 1996-01

CONTACTS AND LOCATIONS:
Overall Officials: William Connor, Study Chair — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States